CLINICAL TRIAL: NCT07364149
Title: Acute Effects of Structured Physical Exercise and Static Passive Stretching on Vascular Function, Neuromuscular Performance, and Metabolic Regulation: A Randomized Crossover Study
Brief Title: Acute Effects of Structured Exercise and Static Stretching on Vascular Function, Neuromuscular Performance, and Metabolic Regulation in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Ewan Thomas, Ewan Thomas, Associate Professor in Psychology, Educational Science and Human Movement, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 353/2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Healthy Participants; Healthy Subjects (HS); Resistance Training Adaptation; Static Stretching; Stretch
Keywords: stretching; static stretching; Resistance training; Resistance exercise; tissue stiffness; blood pressure; Flow Mediated Dilation; heart rate variability; Oxygenation
MeSH Terms: interventions — Resistance Training; Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RT (Experimental): Resistance Training
  Interventions: Other: Resistance Training
- RT+SS (Experimental): Resistance training + Static stretching
  Interventions: Other: Resistance training + Static Stretching
- CC (No Intervention): Control Condition --> participants sat silently on a chair without performing any train

INTERVENTIONS:
Other: Resistance Training — Participants assigned to this group will complete a single supervised upper body resistance training session. The protocol includes bench presses and bicep curls performed at 80% of the individual's 1-rep max, for 4 sets of 8 reps, with standardized rest intervals between sets of 2 minutes. The total duration of the session is approximately 20-30 minutes and does not include any additional static stretching beyond the standardized warm-up.
  Arms: RT
Other: Resistance training + Static Stretching — Participants assigned to this group will complete a single supervised upper body resistance training session. The protocol includes bench presses and bicep curls performed at 80% of the individual's 1-rep max, for 4 sets of 8 reps, with standardized rest intervals between sets of 2 minutes. The total duration of the session is approximately 20-25 minutes .Immediately after the resistance exercises, they will complete a structured static stretching protocol targeting the trained muscle groups (pectoralis and elbow flexors), with each stretch held for about 30 seconds and repeated for several sets. The additional stretching lasts 12 minutes, for a total session duration of about 35-40 minutes.
  Arms: RT+SS

SUMMARY:
This experimental study investigates the acute cardiovascular and vascular responses to a single session of resistance training, with and without additional static stretching, compared with a resting control condition. Participants are allocated to one of three groups (control, resistance training, resistance training plus static stretching) and assessed at baseline, immediately after the session, and 30 minutes post-exercise. Primary outcomes include blood pressure and other hemodynamic or functional measures, in order to explore the short-term impact of these exercise modalities on cardiovascular regulation.

ELIGIBILITY:
Inclusion Criteria:

* healthy male participants ≥ 18 years old

Exclusion Criteria:

* orthopedic disorders
* neurological disorders
* metabolic disorders
* cardovascular disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Dilation(FMD%) | 3 times (Baseline, immediately after intervantion and 30 minutes after intervention) for each condition (CC, RT, RT+ST)
  Brachial artery flow-mediated dilation (FMD) will be assessed using high-resolution B-mode ultrasound (Esaote MyLab X1 GO, linear transducer) during a standardized forearm cuff occlusion protocol. Baseline diameter will be recorded for 60 seconds prior to cuff deflation. Reactive hyperemia will be induced by 5-minutes arterial occlusion followed by cuff release, with continuous diameter recording for 3 minutes post-deflation to identify peak diameter.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No